CLINICAL TRIAL: NCT05908643
Title: A First-In-Human, Phase I/IIa Trial of the Novel T Cell Immunotherapy pTTL in Patients With Advanced Colorectal Cancer
Brief Title: A First-In-Human Trial of pTTL in Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neogap Therapeutics AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry); Karolinska University Hospital (Other); Region Västmanland (Other); Vecura (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neogap-CRC-01
Record Dates: First submitted 2023-03-23; First posted 2023-06-18 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: Immunotherapy; Adoptive cell therapy; T cell therapy; Neoantigens; Autologous cell therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with pTTL (Experimental): A single dose of pTTL will be administered after pre-conditioning chemotherapy with Fludarabine (30 mg/m(2) body surface area) x 3 and Cyclophosphamide (300 mg/m(2) body surface area) x 3 on days -7 to -5. pTTL will usually be infused on day 1 (5 days after last chemotherapy) with the option of administering it on day -3 if judged preferable based on the T cell expansion kinetics during pTTL production. pTTL is administered as a fresh product directly after production.
  Dose escalation will be applied. Cohort 1 (1 patient): 1 million (with an accepted range of down to -5%) viable cells per kg body weight
  Cohort 2 (3 patients): 2.5 million (down to -5%) viable cells per kg body weight
  Cohort 3 (3 patients): 5 million (down to -5%) viable cells per kg body weight
  Cohort 4 (remaining patients): up to 1 billion viable cells
  Interventions: Drug: pTTL

INTERVENTIONS:
Drug: pTTL — pTTL is an autologous cell product for adoptive cancer immunotherapy containing in vitro expanded T cells stimulated with patient-specific tumour neoantigens derived from tumour-draining lymph nodes.
  Other Names: personal tumour-trained lymphocytes

SUMMARY:
This is an open-label, non-randomised FIH trial investigating the safety and tolerability of a novel ATMP, pTTL, composed of autologous tumour-draining lymph node-derived T cells stimulated in vitro with personalised cancer neoantigens.

The neoantigens are selected through a process starting with next generation sequencing (NGS) of tumour material from the patient followed by selection of neoantigenic mutations using an in-house software, PIOR®. Selected neoantigen epitopes are expressed as recombinant proteins, NAG, and used to stimulate T cells to promote neoantigen-specific T cell expansion in vitro in pTTL production.

pTTL is thus based on autologous cells stimulated with patient-specific neoantigens. In consequence, every pTTL product is unique and designated for use in one single individual.

pTTL will be administered to patients with stage IV colorectal cancer (CRC) as a single intravenous dose.

DETAILED DESCRIPTION:
STUDY RATIONALE The present trial is an open-label, non-randomised FIH trial investigating the safety and tolerability of pTTL, an immunotherapy consisting of autologous T cells activated and expanded in vitro using tumour-specific personalised neoantigens. The scientific rationale for pTTL relies on the fact that somatic mutations in tumour cells arising during malignant transformation result in altered proteins or peptides, so called neoantigens. Each individual tumour harbours multiple mutations that form a unique mutation profile, which enables personalisation of each therapeutic product. The neoantigens distinguish tumour cells from normal cells and make the tumour cells targetable by the immune system, and also allows targeting of several targets in the tumour simultaneously. In the present trial, up to 36 neoantigens will be targeted.

The starting material for pTTL is derived from tumour-draining regional lymph nodes (RLNs). The choice of this source of T cells is based on several advantages: The exposure to tumour antigens and, in the case of metastasis, tumour cells causes an enrichment of tumour- specific T cells. These T cells also have the potential to be superior to tumour-infiltrating T cells due to less exposure to tumour-mediated immunosuppression.

The production process for pTTL includes in vitro expansion, which increases the neoantigen-reactive T cell population. The selective T cell expansion is achieved by stimulation with protein constructs containing neoantigen epitopes, based on sequencing data from each patient's own tumour. This improves the chance of effective cancer cell eradication by both increasing the number of cells able to recognise and respond to the tumour, and by breaking immunological tolerance created in vivo by immunosuppressive mechanisms through activation in a non-suppressive environment.

PATIENTS The selected target group of the trial is adults with stage IV CRC. Patients may be considered eligible for inclusion if they have received treatments according to standard of care or if further standard of care treatment options are judged not to be in the patients' best interest (e.g. due to toxicity issues). Patients could also be eligible for inclusion in the trial during a scheduled pause in ongoing palliative therapy, at the discretion of the treating Investigator. Eligible patients must have a primary or metastatic lesion that is accessible to biopsy or surgery to obtain tumour material for NGS analysis. In addition, it is a requirement that the patient can undergo surgical excision of RLNs for use in pTTL production. Eligible patients should also have a good performance status (ECOG 0-1) and organ function, and no pre-existing conditionings deemed to increase their risk for severe side effects of pTTL therapy. Materials for Part I of the trial can be collected, while non-curative therapeutic options remain, and cryopreserved for later use if the patient should become eligible for inclusion in Part II.

METHODOLOGY The trial is composed of 3 parts, referred to as Part I, Part II and Part III.

Patients will be consented separately for Part I and for Part II/III: a first consent is given for tissue collection and pTTL production, and a second consent is given for pTTL treatment, including pre-conditioning chemotherapy and follow-up.

Part I of the trial entails patient identification, recruitment and screening of trial patients. It also comprises production of pTTL, which is performed in 3 steps:

1. Collection of tumour samples and normal samples for NGS and neoantigen selection. Production of stimulatory NAG-coupled beads raw material TC0301.
2. Collection of starting material for pTTL manufacturing from RLN.
3. pTTL manufacturing.

The time required from collection of tumour material and RLNs up until pTTL production and administration to the patient is approximately 8 to 12 weeks. The RLN starting material is cryopreserved after initial processing, enabling flexibility in the timing of pTTL administration.

Part II of the trial entails pre-conditioning and supportive care therapy, treatment with pTTL, and 26 weeks safety follow-up.

Pre-conditioning contains cyclophosphamide and fludarabine, and will be administered between Day -7 and Day -5 before scheduled pTTL administration. Supportive care treatment will start on Day -9 or Day -8. pTTL administration will normally be administered on Day 1, with the option of administration on Day -3 if cell expansion kinetics during pTTL production indicates this would be preferable. Part II will end when the last treated patient has been followed for 26 weeks or earlier in case of death or patient withdrawal.

Part III of the trial is a long-term follow-up initiated after completion of the initial 26 weeks safety follow-up period. Patients will participate in Part III for up to 4.5 years after end of Part II or until death, whichever comes first.

pTTL DOSAGE AND ADMINISTRATION The drug product (DP), i.e. pTTL, is composed of in vitro expanded RLN cells, enriched for neoantigen-specific T cells. It is formulated as a cell suspension with the excipients NaCl (9 mg/mL) and human serum albumin (25 mg/mL) in a transfusion bag intended for intravenous transfusion. The product is administered fresh. Each patient will receive a single administration of pTTL.The cell dose obtained during the manufacturing process will vary depending on the size of the neoantigen-reactive clones present in the starting material and their proliferative capacity. The minimum dose of a pTTL unit is 20 million viable cells and the maximum dose is 1 billion viable cells.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Adult (age ≥18 years).
3. Histological or cytological confirmation of CRC.
4. Verified metastatic disease (stage IV classification) and have received all possible standard of care therapies, OR further standard of care therapies are currently not considered to be in the patient's best interest, OR toxicity from previous therapy limits the choice of suitable standard of care therapy OR scheduled pause in palliative standard of care therapy as judged by the Investigator.
5. Measurable disease according to RECIST1.1.
6. Minimum life expectancy of 6 months at primary inclusion and 3 months at pTTL administration.
7. Minimum life expectancy of 3 months from the time that the individual pTTL DP is estimated to be available (as per Investigators clinical assessment). 7. ECOG performance status 0 to 1
8. Adequate hematopoietic, hepatic and renal function defined as:

   1. Haemoglobin≥ 95 g/L (blood transfusion not less than 21 days prior to screening),
   2. Absolute neutrophil count ≥ 1.0x 109/L, platelets ≥100 x 109/L
   3. Total bilirubin < 1.5 x ULN (does not apply to patients with Gilberts Syndrome)
   4. AST and ALT ≤ 1.5 x ULN (or ≤ 5 x ULN in the presence of liver metastases)
   5. Serum creatinine ≤ ULN (if serum creatinine is between 1 and 1.5 x ULN, patients may be eligible provided that the calculated GFR is at least 35 mL/min using Cockcroft- Gault method).
   6. Albumin ≥24 g/L
9. Patients of childbearing potential or their partners of childbearing potential must be willing to take the appropriate precaution to avoid pregnancy or fathering a child for the duration of Part I and Part II and practice an approved, highly effective method of birth control during treatment and for 6months after receiving pTTL.

   Approved methods of birth control include:
   * Combined (oestrogen and progesterone containing) hormonal birth control associated with inhibition of ovulation: oral, intravaginal, transdermal
   * Progesterone-only hormonal birth control associated with inhibition ofovulation: oral, injectable, implantable
   * Intrauterine device (IUD)or intrauterine hormone-releasing system (IUS)•Bilateral tubal occlusion
   * Vasectomised partner
   * True sexual abstinence when this is in line with the preferred and usuallifestyle of the patient. Periodic abstinence (e.g., calendar ovulation,symptothermal, post-ovulation methods) is not acceptable
10. Able to undergo surgery or biopsy to obtain tumour tissue for neoantigen evaluation and to retrieve RLNs as starting material for pTTL manufacturing
11. The area from which the RLNs will be obtained shall not have been exposed to radiotherapy.

Exclusion Criteria:

1. Less than 4 months at primary inclusion and 6 months at pTTL administration since a clinically significant cardiovascular event such as myocardial infarction, unstable angina, angioplasty, bypass surgery, stroke or transient ischemic attack (TIA). Atrial fibrillation if treated and well controlled is not considered a bar to inclusion even if diagnosed less than 6 months ago.
2. Congestive heart failure New York Heart Association (NYHA)class III or IV.
3. Significantly reduced lung function with clinical implications. If such is suspected, spirometry should be performed. Spirometry should also be considered in patients who have been hospitalised due to Covid-19 infection during the last 6 months, and in patients with any other lung affectation judged significant by the Principal Investigators, in discussion withSponsor's Medical Representative, such as treatment-related pneumonitis or severe lung infection. Spirometry results of less than 65% of the expected value regarding forced expiratory volume in 1 second(FEV1) and/or diffusion capacity (diffusing capacity of the lung for carbon monoxide, DLCO,corrected for haemoglobinvalue, DLCOco) is regarded as a criterium for exclusion.
4. Any severe acute or chronic medical condition that places the patient at increased risk or interferes with the interpretationof trial results (as judged by the Principal Investigators, in agreement with Sponsor's Medical Representative).
5. Immunodeficiency disorders which may pose a risk for patients treated with pTTL, and/or affect the outcome of the pTTL treatment, as judged by Investigator at the Treatment Site and/or the Investigator at the Recruitment and Follow-Up Site Immunodeficiency disorders are here defined as including inborn and acquired disorders reducing immunity but excluding human immunodeficiency virus (HIV), which is discussed below. Examples include common variable immunodeficiency and status post transplantation of a solid organ or stem cells. Immunodeficiency caused by the cancer disorder to be treated within the trial or such cancer treatments as have already been administered is considered a separate entity. This, if severe, might impact the production of pTTL and potentially also the treatment outcome, and needs to be carefully assessed as regards patient and pTTL production risks before inclusion.
6. Autoimmunity disorders which may pose a risk for patients treated with pTTL, and/or affect the outcome of the pTTL treatment, as judged by Investigator at the Treatment Site and/or the Investigator at the Recruitment and Follow-Up Site.
7. Leptomeningeal metastases (patient with previously treated brain metastases are eligible if there is no evidence of disease progression for a minimum of 8 weeks prior to inclusion

   * in these cases a CNS MRI is required within the screening period. These patients must not have symptoms from their brain metastases or treatment thereof and must not be taking steroid medications for treatment of CNS symptoms).
8. Patients are not allowed to have ongoing systemic immunosuppressive concomitant medications. Systemic immunosuppressive treatments should be completed 2 weeks prior to surgery and/or 2 weeks prior to dose. Steroid medications are allowed if they are used as substitution or are administrated topically or as inhalation steroids for asthma.
9. Previous Grade 3 or greater immune-related toxicity from checkpoint modulation or other immunotherapy (unless the toxicity has resolved and the patient rechallenged with the therapy without recurrence of toxicity, in which situation the patient can be considered).
10. Acute or chronic infection with hepatitis B or C or syphilis.
11. HIV infection.
12. Pregnancy or breast-feeding.
13. Investigator considers the patient unlikely to comply with trial procedures, restrictions and requirements.
14. For patients required to undergo trial-specific surgery to obtain starting material:

    1. Less than 3 identifiable enlarged lymph nodes on pre-surgery radiology accessible for surgical excision.
    2. Previous surgical removal of the primary CRC tumour (would entail a high risk surgery)
    3. Unable to withstand the planned surgery (including ineligibility for general anaesthesia)

    At decision to proceed to pTTL administration:
15. Less than 4 weeks since stopping previous systemic cancer treatment.
16. Less than 2 weeks since stopping radiotherapy.
17. Less than 4 weeks after major surgery and less than 3 weeks after minor surgery.
18. Participation in any other clinical cancer therapy trial, and planned treatment or treatment with another investigational drug, within the previous 4 weeks.
19. Less than 4 weeks since administration of live attenuated vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Safety of pTTL administration, as determined by assessment of incidence and severity of adverse events (AE). Immunological AEs and AEs known to be associated with T cell therapies will be classified as AEs of special interest (AESI). | Final evaluation 6 months after pTTL therapy
  To establish that pTTL can be administered to patients with advanced CRC without unacceptable toxicity. Adverse events (AEs) will be collected and assessed according to Common terminology criteria for AEs (CTCAE) v5.0. Special focus will be placed on immunological AEs and AEs known to be associated with T cell therapies, defined as AEs of special interest (AESI). AESI will include autoimmune reactions potentially resulting from off-target toxicity such as colitis, and immune-mediated reactions associated with immune cell activation, such as cytokine release syndrome (CRS).

SECONDARY OUTCOMES:
Objective response | Final evaluation 6 months after pTTL therapy
  Measured using radiology (including CT, MR or other applicable examination) and assessed according to iRECIST
Time to treatment response | Final evaluation 6 months after pTTL therapy
  The time between administration and documented objective response
Duration of treatment response | Final evaluation 6 months after pTTL therapy
  The time from when an objective response is initially documented to the time of subsequent tumour progression.
Time to tumour progression | Final evaluation 6 months after pTTL therapy
  The time to tumour progression after pTTL administration will be assessed using the iRECIST criteria and will take into account the time from inclusion in Part II of the trial until disease progression.
Kinetics of tumour progression/growth (compared to pre-treatment) | Final evaluation 6 months after pTTL therapy
  This measurement will be based on iRECIST, and will use radiological examinations (including CT, MR or other applicable examination) before and after pTTL administration in an endeavour to evaluate whether the progression kinetics of the patient's cancer is affected by pTTL administration
Overall survival | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Defined as time from inclusion to death of any cause.
Progression-free survival | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Defined as time from inclusion to tumour progression or death of any cause.
Disease-specific survival | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Defined as time from inclusion to death of disease.

OTHER OUTCOMES:
Biomarker analysis for evaluation of pTTL persistence | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  T cell receptor sequencing (TCRseq) will be used to characterise the pTTL product and to trace the identified pTTL clones in sequential peripheral blood samples post treatment.
Biomarker analysis for evaluation of pTTL tumour infiltration | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  If feasible, pre- and post-treatment biopsies will be taken for histological assessment of T cell infiltration and characterisation of tumour-infiltrating T cells.
Biomarker analysis for evaluation of pTTL neoantigen specificity | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Functional T cell assays (including but not limited to flow cytometry and cytokine release assays) will be used to evaluate neoantigen-specific responses in the pTTL product and in peripheral blood T cells, reflecting the extent of neoantigen reactivity in the different samples.
Biomarker analysis for evaluation of pTTL neoantigen efficacy - serum tumour markers | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Serum tumour markers (the choice of markers will be made according to the patient's tumour characteristics) will be assessed as a biomarker of efficacy, as it reflects changes in tumour burden.
Biomarker analysis for evaluation of pTTL neoantigen efficacy - ctDNA | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Circulating tumour DNA (ctDNA) will be assessed as a biomarker of efficacy, as it reflects changes in tumour burden.
Biomarker analysis for evaluation of pTTL characteristics | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Analysis of the pTTL product and of post therapy peripheral blood samples will be performed to evaluate the functional status, differentiation and lineage-identity of T cells and other immune cells. This is an exploratory outcome measure, where a large set of phenotypical aspects will be assessed in order to understand which characteristics are important for pTTL efficacy and potentially also to side effects. Evaluations of the T cells are performed using assays including, but not limited to, flow cytometry and RNA sequencing, to characterize the T cells with regard to identity, differentiation and functions which could be relevant to the efficacy of pTTL.
Evaluation of the importance of neoantigen selection to clinical outcome. | First evaluation at 6 months after pTTL therapy, with a final evaluation at the close of the study at a maximum of 5 years after pTTL administration.
  Data relevant for the correlation of neoantigen selection to clinical outcome will be stored and assessed. Aspects such as type of genetic alteration, variant allele frequency, RNA expression, and protein type and function will be considered and assessed in the context of clinical outcomes, signals of efficacy and biomarker evaluation. This is an exploratory outcome measure, and multiple assessments will be performed to better understand what neoantigen characteristics that could affect efficacy of pTTL.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Kordes, MD, PhD, Principal Investigator — Medical Unit Cell therapy and Allogeneic Stem cell Transplantation, Karolinska University Hospital; Abbas Chabok, MD, PhD, Principal Investigator — Unit for Colorectal Surgery, Dept. of Surgery, Västmanlands Sjukhus Västerås
Locations (2):
- Sweden (2):
  - Medical Unit Cell therapy and Allogeneic Stem cell Transplantation (ME CAST), and the Center for Clinical Cancer studies - Phase 1 unit, Karolinska University Hospital, Stockholm, Stockholm County
  - Unit for Colorectal Surgery, Dept. of Surgery, Västmanlands Sjukhus Västerås, Västerås, Västerås